CLINICAL TRIAL: NCT05185180
Title: Effects of Epigenetic Regulation in Chronic Pelvic Pain Syndrome
Status: Active, not recruiting | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Praveen Thumbikat, O'Connor Family Research Professor of Urology, Northwestern University
Other Study IDs: STU00215831
Record Dates: First submitted 2021-11-05; First posted 2022-01-11 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Chronic Pelvic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — * Undergo specimen collection of:
    * Void Bladder 1, 2, and 3 (10mL of urine, each; 30mL total)
    * Expressed prostatic secretion (EPS)
    * Peripheral blood (3 tubes, 10mL each)
  * Complete baseline questionnaires
    * National Institutes of Health Chronic Prostatitis Symptom Index (NIH-CPSI)
    * American Urological Symptom Index (AUA-SI)
  * A Physical examination including vital heart rate, breathing rate, blood pressure, temperature, height, weight and body mass will be taken
  * Provide a basic health history, including current general health, adverse events, medications or treatments within the past 5 years.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Males with Category III Chronic Pelvic Pain Syndrome: Category III is subdivided into inflammatory (IIIa) and noninflammatory (IIIb) subtypes, based on the presence of white blood cells in expressed prostatic secretions (EPS). Category III prostatitis or chronic pelvic pain syndrome (CPPS) is the most common prostatitis observed in medical practice with a prevalence rate in the general population from 5% to 14.2%. CPPS is a poorly understood entity characterized by pelvic or perineal pain, irritative voiding symptoms, and sexual dysfunction.
- Control Group: The control group will consist of men with no history of Chronic Pelvic Pain or any underlying condition.

SUMMARY:
This study seeks to identify defects in immune activation or regulation that may affect a subset of patients with CP/CPPS. This subset appears to have a reduced ability to mount a regulatory immune response, while simultaneously eliciting an exaggerated activated immune response. The defects that we demonstrate appear to be linked to altered methylation of genes involved in both immune regulation and immune activation. The aims of this study will provide definitive evidence of a role for epigenetic changes in immune cells in patients with CP/CPPS.

DETAILED DESCRIPTION:
CPPS is a condition that is estimated to affect up to 15% of the male population with most diagnoses between the ages of 35-45. Designated by the presence of pain in the absence of bacterial infection for more than three months, it has unknown, probably complex etiology, which thus far have hampered efforts to determine effective treatment strategies. The heterogeneous nature of the symptoms and the length of the disease course prior to detection, presentation or diagnosis only further exacerbate these issues. This study seeks to identify defects in immune activation or regulation that may affect a subset of patients with CP/CPPS. This subset appears to have a reduced ability to mount a regulatory immune response, while simultaneously eliciting an exaggerated activated immune response. The defects that we demonstrate appear to be linked to altered methylation of genes involved in both immune regulation and immune activation. The aims of this study will provide definitive evidence of a role for epigenetic changes in immune cells in patients with CP/CPPS. This is conceptually a major advance - as a variety of factors including early life stress events, prostate infectious agents, environmental variables, all could contribute to epigenetic change and may therefore explain both the anecdotal etiologies described in this syndrome as well as the difficulty in pinpointing a precise etiological mechanism. Specifically, our data leads us to hypothesize that epigenetic alterations in regulatory and proinflammatory immune pathways underpin the development of chronic pelvic pain in CPPS. In this study, we propose to validate our preliminary findings in a larger set of CP/CPPS patients and controls as well as utilize murine models of prostatitis to understand the mechanism driving altered IL-10 and IL-7/LFA-1 mediated immune responses both at systemic and prostate levels. If epigenetic defects and functional deficits can be demonstrated, diagnosis and treatment methodologies could be better targeted at correction of these chronic deficits rather than at etiological agents/pathways that are in the past.

BACKGROUND:

Prostatitis accounts for approximately 2 million outpatient visits per year in the United States, including 1% of those to primary care physicians. Chronic pelvic pain syndrome (CPPS) accounts for 90% of all chronic prostatitis but has no well-defined etiology. It is clinically characterized by the symptoms of pain in the perineum, testes, penis, suprapubic area, dysuria and profound reductions in patient quality of life. Epidemiologic observations indicate that prostatitis conditions are the most frequent urologic diagnosis in young men and the third most frequent urologic diagnosis in men older than 50 yr, representing 8-12% of urology office visits. The NIH consensus definition and classification identifies four categories of prostatitis. Categories I and II have bacterial etiologies while the rest are believed to be non- bacterial in etiology.

Category III is subdivided into inflammatory (IIIa) and noninflammatory (IIIb) subtypes, based on the presence of white blood cells in expressed prostatic secretions (EPS). Category III prostatitis or chronic pelvic pain syndrome (CPPS) is the most common prostatitis observed in medical practice with a prevalence rate in the general population from 5% to 14.2%. CPPS is a poorly understood entity characterized by pelvic or perineal pain, irritative voiding symptoms, and sexual dysfunction.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Control Group:

• Healthy males ages 21-80 years old

Exclusion Criteria:

Exclusion Criteria for Control Group:

* Females
* Males <21 and >80 years old
* Patients with impaired renal or hepatic function.

Ages: 21 Years to 80 Years | Sex: Male
Age Groups: Adult, Older Adult
Gender Based: Yes — Recruiting healthy males with no history of chronic pelvic pain or no underlying conditions to be the control group for effects of epigenetic regulation in chronic pelvic pain syndrome
Study Population: We hypothesize that aberrant immune regulation and/or activation due to epigenetic alterations in immune genes facilitate chronic pelvic pain. The objective of this aim is to expand on our preliminary data demonstrating epigenetic modifications in immune-related genes in CP/CPPS patients compared to healthy controls. To do so, we propose to recruit CP/CPPS patients and healthy volunteers to obtain peripheral blood and prostate secretions (EPS) for performing tailored methylation arrays on PBMC's, examination of functional consequences of immune alterations and finally correlation with patient symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-10-11 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12-11 (Estimated)

PRIMARY OUTCOMES:
Identifying immune-related epigenetic modifications in patients with CP/CPPS. | 5 Years
  To recruit CP/CPPS patients and healthy volunteers to obtain peripheral blood and prostate secretions (EPS) for performing epigenetic analysis of PBMC
Identifying immune-related modifications in patients with CP/CPPS. | 5 Years
  To recruit CP/CPPS patients and healthy volunteers to obtain peripheral blood and prostate secretions (EPS) for examination of immune changes.
Identifying patient symptoms in CP/CPPS. | 5 Years
  To recruit CP/CPPS patients and healthy volunteers to obtain peripheral blood and prostate secretions (EPS) for examining correlation with patient symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Praveen Thumbikat, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States